CLINICAL TRIAL: NCT05754658
Title: African Cancer Genome Cohort to Promote Health Equity Among Patients of African Ancestry: Characterization of Genetic and Molecular Drivers
Brief Title: African Cancer Genome: GMD
Status: Recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: University of Miami Sylvester Comprehensive Cancer Center (Other); Pfizer (Industry); The University of The West Indies, Mona, Jamaica (Unknown); Kenya Medical Research Institute (Other); University of Nairobi, Kenya (Unknown); University of Abomey Calavi, Benin (Unknown); Innovating Health International, Haiti (Unknown); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); The University of the West Indies at Cave Hill, Barbados (Unknown); The University of The West Indies School of Clinical Medicine and Research, The Bahamas (Unknown); Ministry of Health and Social Services, Namibia (Other Government); Morgan State University (Other); University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Camille Ragin, PhD, MPH, Professor, Fox Chase Cancer Center
Other Study IDs: 22-4004
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and FFPE samples for DNA and RNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Cancer: Female patients
  Interventions: Other: Standard of Care
- Prostate Cancer: Male patients
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Drugs routinely administered for breast cancer per local standard.
  Groups: Breast Cancer
Other: Standard of Care — Drugs routinely administered for prostate cancer per local standard.
  Groups: Prostate Cancer

SUMMARY:
The goal of this study is to develop a comprehensive characterization of genetic and molecular drivers of breast and prostate cancer in individuals of African ancestry. The study is conducted by the African Caribbean Cancer Consortium (AC3) and involves the recruitment of patients from nine international AC3 research sites in the Bahamas, Barbados, Benin, Burkina Faso, Haiti, Jamaica, Kenya, Namibia, and Trinidad and Tobago, and the US. The main questions are to: molecularly characterize genomic changes in the African Cancer genomes of the breast and prostate and identify the effects of social determinants of health and lifestyle factors on mutational landscape. Black individuals that have been diagnosed with pathologically confirmed prostate or breast cancer will be included. Detailed social determinants of health survey, blood and archived FFPE tissues will be collected. (Tier 1) All patient tissues will be subject to IHC for receptor status (ER, AR, PR Her2/neu). All patients with available germline DNA from blood will receive genetic screening using a Commercial gene panel testing. (Tier 2) Patient samples with a negative genetic screening will be subject to whole exome sequencing or banked for later RNA or methylation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18-85 years of age, diagnosed with a pathologically confirmed cancer at any stage at diagnosis. Participant can have a history of a previous cancer we will control for previous history of cancer diagnosis in our analysis.

Exclusion Criteria:

* Patients age <18 year, incarcerated patients, and patients whose medical decisions are made by proxy will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females who self-identify as Black with a pathologically confirmed diagnosis of prostate or breast cancer are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemistry | Year 1-2
  ER, PR, Her2 and AR status in breast and prostate tissues
Germline Mutations | Year 1-2
  Hereditary mutations in germline DND from breast and prostate
Mutational Landscape | Year 2
  tumor mutation burden in breast and prostate tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States